CLINICAL TRIAL: NCT07393802
Title: Evaluation of the Anti-Plaque Effect of a Resveratrol-Based Mouthwash Using a 24-Hour Plaque Biofilm Re-Growth Randomized Crossover Clinical Trial
Brief Title: Evaluation of the Anti-Plaque Effect of a Resveratrol-Based Mouthwash Using a 24-Hour Plaque Re-Growth
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Ahmed Hashim Alyasari, Assistant professor of periodontology, University of Baghdad
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 07731873348
Record Dates: First submitted 2026-01-22; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Mouthwash; Chlorhexidine; Biofilm Formation; Periodontal Health
Keywords: Resveratrol; mouthwash; anti-plaque; crossover
MeSH Terms: interventions — chlorhexidine gluconate; Mouthwashes

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The products will be packaged in such a way that they are not recognizable neither by the operator, nor by the patient. Each package will be assigned a number that in turn will refer to the type of the product. The association between the number and type of the product will be collected by another operator according to the association carried out by a dedicated software. The operator who will deliver the product will be informed about the type only at the end of the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resveratrol-Based Mouthwash (Experimental): Participants assigned to this arm will rinse with 10 mL of the resveratrol-based mouthwash for 30 seconds. Following rinsing, participants will be instructed to refrain from eating or drinking for at least 30 minutes.
  The mouthwash will be used twice daily (at baseline and after 12 hours). During the 24-hour plaque re-growth period, participants will be instructed to avoid all forms of mechanical oral hygiene, including toothbrushing, flossing, and the use of any additional oral hygiene products.
  Interventions: Drug: Resveratrol-Based Mouthwash
- Chlorhexidine Mouthwash (0.12%) (Active Comparator): Participants assigned to this arm will rinse with 10 mL of 0.12% chlorhexidine digluconate mouthwash for 30 seconds. After rinsing, participants will be instructed to refrain from eating or drinking for at least 30 minutes.
  The mouthwash will be used twice daily (at baseline and after 12 hours). Throughout the 24-hour plaque re-growth period, participants will be instructed to avoid all mechanical oral hygiene measures, including toothbrushing, flossing, and the use of any additional plaque control products.
  Interventions: Drug: Chlorhexidine Gluconate 0.12 % Mouthwash
- Placebo mouthwash (Placebo Comparator): Participants assigned to this arm will rinse with 10 mL of a placebo mouthwash for 30 seconds. After rinsing, participants will be instructed to refrain from eating or drinking for at least 30 minutes.
  The mouthwash will be used twice daily (at baseline and after 12 hours). During the 24-hour plaque re-growth period, participants will be instructed to avoid all mechanical oral hygiene measures, including toothbrushing, flossing, and the use of any additional oral hygiene products.
  Interventions: Drug: Placebo mouthwash

INTERVENTIONS:
Drug: Resveratrol-Based Mouthwash — This intervention represents the test group of the study and consists of a resveratrol-based mouthwash (Oroxil®), a patented formulation containing resveratrol and carvacrol. The mouthwash is evaluated as a chemical plaque control agent to assess its short-term anti-plaque efficacy using a 24-hour supragingival plaque re-growth model. The intervention is administered under controlled clinical conditions and compared with chlorhexidine and placebo mouthwashes within a randomized, double-blind, crossover study design.
  Arms: Resveratrol-Based Mouthwash
Drug: Chlorhexidine Gluconate 0.12 % Mouthwash — This intervention represents the positive control group of the study and involves the use of a 0.12% chlorhexidine digluconate mouthwash. The mouthwash is employed as a reference chemical plaque control agent to evaluate its short-term anti-plaque effect using a 24-hour supragingival plaque biofilm re-growth model. The intervention is administered under standardized and controlled clinical conditions and is compared with the resveratrol-based mouthwash and a placebo within a randomized, double-blind, three-period crossover study design.
  Arms: Chlorhexidine Mouthwash (0.12%)
Drug: Placebo mouthwash — This intervention represents the negative control group of the study and involves the use of a placebo mouthwash with no active antimicrobial ingredients. The placebo is used to assess supragingival plaque biofilm re-growth under standardized conditions and to provide a baseline comparison for evaluating the short-term anti-plaque effects of the resveratrol-based and chlorhexidine mouthwashes. The intervention is administered under controlled clinical conditions within a randomized, double-blind, three-period crossover study design.
  Arms: Placebo mouthwash

SUMMARY:
Dental plaque is a biofilm that accumulates on tooth surfaces and is a primary factor in the development of gingival inflammation. While toothbrushing remains the main method for plaque control, the effectiveness of mechanical oral hygiene depends largely on individual compliance and technique. As a result, mouthwashes are commonly used as adjunctive chemical plaque control agents.

Chlorhexidine gluconate is an effective anti-plaque mouthwash, but its use is associated with undesirable effects that may limit patient acceptance. Resveratrol is a naturally derived compound with reported antimicrobial and anti-biofilm properties, suggesting its potential use as an alternative chemical plaque control agent.

This randomized, double-blind, placebo-controlled, three-period crossover clinical trial aims to evaluate the short-term anti-plaque effect of a resveratrol-based mouthwash by measuring supragingival plaque regrowth over a 24-hour period in periodontally healthy individuals. The effects of the resveratrol-based mouthwash will be compared with 0.12% chlorhexidine (CHX) and a placebo mouthwash under standardized conditions without mechanical oral hygiene

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, three-period crossover clinical trial conducted in periodontally healthy individuals to evaluate the short-term anti-plaque efficacy of a resveratrol-based mouthwash. The study population will consist of systemically healthy undergraduate dental students with clinically healthy gingiva and no signs of gingivitis or periodontitis. This population was selected to allow accurate assessment of supragingival plaque re-growth without the influence of periodontal inflammation or periodontal pocketing.

Prior to the clinical trial, participants will undergo a one-week preparatory period during which oral hygiene instructions will be provided and professional scaling and polishing will be performed to obtain plaque-free tooth surfaces. Standardized oral hygiene aids will be supplied for use during the preparatory and washout periods.

Participants will be randomly assigned to different intervention sequences determining the order of the three mouthwashes using a computer-generated randomization list prepared by an independent individual not involved in the clinical examinations. To minimize bias, the study will be conducted in a double-blind manner, with the test, positive control, and placebo mouthwashes dispensed in identical opaque bottles. Both participants and the examiner will remain blinded to the identity of the interventions until completion of all study phases.

At the beginning of each intervention period, supragingival plaque will be disclosed and removed by professional polishing to standardize baseline conditions. Participants will then rinse with 10 milliliters of the assigned mouthwash for 30 seconds under supervision and will be instructed to refrain from eating or drinking for 30 minutes. A second rinse will be performed after 12 hours. Participants will be instructed to refrain from all mechanical oral hygiene measures and the use of additional oral hygiene products during the 24-hour experimental period.

After 24 hours, supragingival plaque accumulation will be assessed using the Modified Quigley-Hein Plaque Index (MQHPI). Digital plaque image analysis (DPIA) will be performed using fluorescein-disclosed ultraviolet images to quantify plaque-covered tooth surfaces. Following plaque assessment, professional polishing will be carried out.

Each intervention phase will be separated by a six-day washout period to minimize potential carryover effects. During the washout period, participants will resume routine oral hygiene practices using standardized oral hygiene aids. The short-term safety and acceptability of the tested mouthwashes will be assessed throughout the study

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 30 years
* Systemically healthy individuals
* Presence of at least 20 natural teeth
* Clinically healthy gingiva with no signs of gingivitis or periodontitis
* No probing depth >3 mm
* No clinical attachment loss

Exclusion Criteria:

* Presence of gingivitis or periodontitis
* Active dental caries requiring treatment
* History of periodontal therapy within the previous 6 months
* Use of antibiotics, anti-inflammatory drugs, or antiseptic mouthwashes within the previous 3 months
* Smoking or tobacco use
* Pregnancy or lactation
* Known allergy to any mouthwash components

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Supragingival Plaque Accumulation Assessed by the Modified Quigley-Hein Plaque Index (MQHPI) | 24 hours
  Supragingival plaque accumulation will be assessed after 24 hours using the MQHPI. Plaque scores will be recorded for each participant and used to compare plaque accumulation between the different mouthwash interventions.

SECONDARY OUTCOMES:
Percentage of Plaque-Covered Tooth Surface Assessed by Digital Plaque Image Analysis (DPIA) | 24 hours
  Plaque coverage will be assessed after 24 hours using the DPIA. Fluorescein-disclosed plaque images will be obtained, and the percentage of plaque-covered tooth surface will be calculated by dividing the number of pixels classified as plaque on teeth by the total number of pixels representing plaque and tooth surfaces, multiplied by 100. The resulting percentage values will be used for comparison between the different mouthwash interventions
Number of Participants With Oral Adverse Effects Related to Mouthwash Use | 24 hours
  The number of participants experiencing treatment-related oral adverse effects, including oral irritation, burning sensation, mucosal changes, or discomfort, will be assessed during and after each 24-hour intervention period based on clinical examination and participant report.
Participant-Reported Taste Acceptability of the Tested Mouthwashes | 24 hours
  Taste acceptability of each mouthwash will be assessed after each 24-hour intervention period using participant self-report.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Hashim, Karbala, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mohammed SA, Akram HM. Evaluating the Efficacy of Resveratrol-Containing Mouthwash as an Adjunct Treatment for Periodontitis: A Randomized Clinical Trial. Eur J Dent. 2025 May;19(2):354-365. doi: 10.1055/s-0044-1788686. Epub 2024 Sep 9. PMID 39251207
- [Result] Abed Taher NA, Mahmood AA, Hussein HM. Efficacy of a Mouthwash Containing Resveratrol in Reducing Halitosis-related P. gingivalis: A Randomized Triple-blind Trial. Oral Health Prev Dent. 2025 Dec 2;23:793-803. doi: 10.3290/j.ohpd.c_2373. PMID 41328922